CLINICAL TRIAL: NCT04044742
Title: A Phase 3 Placebo-controlled Study to Evaluate the Efficacy and Safety of Intra-articular Administration of Resiniferatoxin Versus Placebo for the Treatment of Moderate to Severe Pain Due to Osteoarthritis of the Knee
Brief Title: A Phase 3 Study to Evaluate the Efficacy and Safety of Resiniferatoxin for Pain Due to Osteoarthritis of the Knee
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: To be replaced by a different protocol
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STI-RTX-3001
Record Dates: First submitted 2019-08-02; First posted 2019-08-05 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Osteoarthritis, Knee; Knee Pain Chronic
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — resiniferatoxin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The treatment assigned to each subject is blinded to the subject, investigators, and sponsor study team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resiniferatoxin (Experimental): 12.5 ug of Resiniferatoxin in 5 mL volume is administered as a one-time dose, intra-articularly
  Interventions: Drug: Resiniferatoxin
- Placebo (Placebo Comparator): Placebo formulation in 5 mL volume administered intra-articularly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Resiniferatoxin — Receiving Resiniferatoxin injection
  Other Names: RTX
  Arms: Resiniferatoxin
Drug: Placebo — Receiving Placebo injection
  Other Names: Diluent
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy and safety of intra-articular injection of resiniferatoxin in patients with moderate to severe knee pain due to osteoarthritis.

DETAILED DESCRIPTION:
This study is to evaluate the analgesic efficacy and safety of resiniferatoxin administered intra-articularly to subjects with moderate to severe knee pain due to osteoarthritis (OA).

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female 35 to 85 years of age (inclusive).
* Diagnosis of moderate to severe pain in the index knee due to OA.
* Pain in the non-index knee is less than pain in the index knee.
* Body mass index ≤40 kg/m².
* Experienced treatment failure with at least 2 prior categories of therapies.
* Able to understand and complete study-related forms and communicate with the Investigator and/or site staff.

Key Exclusion Criteria:

* Evidence or history of a serious coagulopathy or hemostasis problem, such as inherited bleeding disorders or thrombocytopenia.
* History of or current condition of poorly controlled hypertension, QTc prolongation, history of risk factors for Torsades de Pointes, or family history of long QT syndrome; or is using concomitant medications that prolong the QT interval.
* Received index knee injections with corticosteroids within 30 days, or hyaluronic acid within 3 months, or platelet-rich plasma within 6 months prior to the injection day.
* Pre-existing osteonecrosis, subchondral insufficiency fracture, severe bone on bone OA, or knee pain attributable to disease other than OA.
* Instability or misalignment in the index knee.
* Concurrent use of opioids or indications other than knee pain.
* History within the past 2 years of substance abuse, including alcohol.
* Allergy or hypersensitivity to chili peppers, capsaicin, resiniferatoxin, acetaminophen, tramadol, or radiographic contrast agents.
* Female participants who are pregnant, planning on becoming pregnant, or currently breastfeeding.
* Any medical condition or comorbidities that, in the Investigator's opinion, could adversely impact study participation or safety, conduct of the study, or interfere with pain assessments.
* Sensory peripheral neuropathy that is of moderate severity or higher.
* Arterial or venous thrombi (including stroke), myocardial infarction, hospital admission for unstable angina, cardiac angioplasty, or stenting within the past 12 months.
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome-related illness, acute or history of chronic hepatitis B or hepatitis C. Participants with these viral infections who are receiving or have received antiviral treatment and have a viral load that is undetectable are eligible.
* Concurrent medical or arthritic conditions that could interfere with the evaluation of the index knee joint including chondromalacia patellae, metabolic diseases, gout/pseudogout, hemochromatosis, acromegaly, fibromyalgia, rheumatoid arthritis, or other inflammatory arthropathies affecting the knee joint.
* Undergone arthroscopic surgery of the index knee within 6 months of the injection day, or open surgery to the index knee within 24 months of the injection day.
* Undergone replacement surgery of the index knee.
* Presence of surgical hardware or other foreign bodies in the index knee.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change in index knee pain with walking | Baseline through Week 12
  Change in the weekly mean of Average Daily Pain (ADP) scores in the index knee, using the 10-point Numerical Pain Rating Scale (NPRS)

SECONDARY OUTCOMES:
Area under the curve (AUC) change in average pain in the index knee | Baseline through Week 12
  AUC calculated on change in the average pain in the index knee over the previous 24 hours, using the NPRS (0-10)
Change in index knee pain with walking | Baseline through Week 26
  Change in the weekly mean of ADP scores in the index knee, using the NPRS (0-10)
AUC change in average pain in the index knee | Baseline through Week 26
  AUC calculated on change in the average pain in the index knee over the previous 24 hours, using the NPRS (0-10)
Duration of effect of a single injection in the index knee | Baseline through return to Baseline
  Time to return to baseline pain score, based on weekly average NPRS (0-10) scores
Change in index knee pain, stiffness, and physical function | Baseline through Week 12, Week 26, and Week 52
  Change in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) total score
Change in the average pain in the index knee | Baseline through Week 12, Week 26, and Week 52
  Change in the WOMAC A pain subscale
Change in the average stiffness in the index knee | Baseline through Week 12, Week 26, and Week 52
  Change in the WOMAC B function subscale
Change in the average function in the index knee | Baseline through Week 12, Week 26, and Week 52
  Change in the WOMAC C stiffness subscale
Change in index knee pain with walking | Baseline through Week 52
  Change in the weekly mean of ADP scores in the index knee, using the NPRS (0-10)
AUC change in average pain in the index knee | Baseline through Week 52
  AUC calculated on change in the average pain in the index knee over the previous 24 hours, using the NPRS (0-10)
Change in quality of life (QOL) - SF-36 Health Survey | Baseline through Week 12, Week 26, and Week 52
  Change in QOL as measured by the SF-36 Health Survey
Change in quality of sleep | Baseline through Week 12, Week 26, and Week 52
  Change in quality of sleep as measured by the MOS Sleep Scale
Patient Global Impression of Change | At Week 12, Week 26, and Week 52
  Rating of change in index knee pain using the PGIC scale
Change in QOL - EQ-5D-5L | Baseline through Week 12, Week 26, and Week 52
  Change in QOL as measured by the EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Monica Luchi, MD, Study Director — Sorrento Therapeutics, Inc.

IPD SHARING:
Plan to Share IPD: No